CLINICAL TRIAL: NCT02892344
Title: A Multi-center, Randomized, 12-week Treatment, Doubleblind Study to Assess the Efficacy and Safety of QMF149 (150/80 Microgram) Compared With MF Twisthaler® (200 Microgram) in Adult and Adolescent Patients With Asthma
Brief Title: Study of QMF149 (150/80 µg) Compared With MF Twisthaler® (200 µg) in Patients With Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CQVM149B2303; 2016-000472-22 (EudraCT Number)
Record Dates: First submitted 2016-08-29; First posted 2016-09-08 (Estimated); Results first posted 2019-09-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Mild Asthma
Keywords: Phase III, blinded, QMF149, Mometasone furoate (MF), mild asthma, Adolescent, adult
MeSH Terms: interventions — QMF149; indacaterol; Mometasone Furoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- QMF149 150/80 μg (Experimental): QMF149 150/80 microgram o.d. delivered via Concept1
  Interventions: Drug: QMF149 150/80 μg
- MF 200 µg (Active Comparator): MF 200 microgram o.d. delivered via Twisthaler®
  Interventions: Drug: MF 200 μg

INTERVENTIONS:
Drug: QMF149 150/80 μg — QMF149 150/80 μg o.d via Concept1
  Other Names: Indacaterol acetate/Mometasone furoate
  Arms: QMF149 150/80 μg
Drug: MF 200 μg — MF 200 μg o.d. via Twisthaler®
  Other Names: Mometasone furoate
  Arms: MF 200 µg

SUMMARY:
The purpose of the trial was to evaluate efficacy and safety of QMF149 150/80 microgram o.d.

delivered via Concept1 compared to MF 200 microgram o.d., delivered via Twisthaler® in terms of lung function and symptom control in poorly (ie inadequately) controlled asthma patients. This study was to assess contribution of LABA as an add-on therapy to low dose ICS monotherapy.

DETAILED DESCRIPTION:
The primary objective of this study was to demonstrate the superiority of QMF149 150/80 microgram o.d. (in the evening) delivered via Concept1 compared with MF 200 microgram o.d. (in the evening) delivered via Twisthaler® in terms of trough FEV1 after 12 weeks of treatment in adults and adolescents. The key secondary objective of this study was to demonstrate the superiority of QMF149 150/80 microgram to MF 200 microgram o.d. in terms of ACQ-7 after 12 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a documented diagnosis of asthma for a period of at least 3 months prior to Screening Visit
* Patients who have used low dose ICS , with or without controller (ie, LABA, Leukotriene Receptor Antagonist ) at stable dose for at least 1 month prior to Screening Visit
* Adult patients who are symptomatic at screening despite treatment with existing therapy.

Patients with ACQ-7 score ≥ 1.5 at Visit 101 and at Visit 102 (inadequately controlled).

* Adolescent patients :
* If taking only ICS (without LABA) and are symptomatic at screening despite treatment with low doses of ICS. These patients must have ACQ-7 score ≥ 1.5 at Visit 101 and at Visit 102 .
* If taking ICS (low dose)/ LABA, and have ACQ-7 score ≥1 and <1.5 at Visit 101: they must have ACQ-7 score≥1.5 at Visit 102 ( prior to randomization).
* Pre-bronchodilator FEV1≥ 60 % and < 90 % of the predicted normal value for the patient after withholding bronchodilators at both Visits 101 and 102
* Patients who demonstrate an increase in FEV1 of 12% and ≥ 200 mL within 30 minutes after administration of 400 microgram salbutamol/360 microgram albuterol (or equivalent dose) at Visit 101.

Exclusion Criteria:

* Patients who have smoked or inhaled tobacco products (including electronic cigarettes) within the 6 month period prior to Visit 1, or who have a smoking history of greater than or equal to 10 pack year.
* Patients who have had an asthma attack/exacerbation requiring systemic steroids or hospitalization (> 24 hours) or emergency room visit (≤ 24 hours) as follows:
* For adults: within 6 weeks of Screening Visit. If patients experience an asthma attack/exacerbation requiring systemic steroids or emergency room visit between Visit 1 and Visit 102 they may be re-screened 6 weeks after recovery from the exacerbation
* For adolescents: Severe asthma attack/exacerbation requiring systemic corticosteroids in the last 6 months, OR hospitalization (> 24 hours) due to severe asthma attack/exacerbation requiring systemic corticosteroids in the last 6 months, OR emergency room visit (≤ 24 hours) due to severe asthma attack/exacerbation requiring systemic corticosteroids within the last 6 months.
* Patients who ever required intubation for a severe asthma attack/exacerbation
* Patients with a clinical condition (eg. glaucoma, cataract and fragility fractures) which may be worsened by ICS administration (according to investigator's medical judgment )
* Patients who have had a respiratory tract infection or asthma worsening within 4 weeks prior to Screening Visit or between Visit 1and Visit 102. Patients may be re-screened 4 weeks after recovery from their respiratory tract infection or asthma worsening.
* Patients with any chronic conditions affecting the upper respiratory tract (eg. chronic sinusitis) which in the opinion of the investigator may interfere with the study.
* Patients with a history of chronic lung diseases other than asthma, including (but not limited to) COPD, sarcoidosis, interstitial lung disease, cystic fibrosis, clinically significant bronchiectasis and active tuberculosis.
* Patients with Type I diabetes or uncontrolled Type II diabetes.
* Patients with narcolepsy and/or insomnia.
* Patients on Maintenance Immunotherapy (desensitization) for allergies or less than 3 months prior to Visit 101 or patients on Maintenance Immunotherapy for more than 3 months prior to Visit 101 but expected to change throughout the course of the study.
* Patients with diagnosed rare hereditary problems of galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption or with known intolerance to lactose or milk products.

  * Patients who use a long acting muscarinic antagonist (LAMA) within 3 months prior to Visit 1.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 802 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2018-11-05 (Actual); Study Completion 2018-11-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (116):
- Bulgaria (3):
  - Novartis Investigative Site, Bulgaria, Bulgaria
  - Novartis Investigative Site, Stara Zagora, Bulgaria
  - Novartis Investigative Site, Pleven
- Chile (3):
  - Novartis Investigative Site, Santiago, Santiago Metropolitan
  - Novartis Investigative Site, Santiago
  - Novartis Investigative Site, Viña del Mar
- Colombia (5):
  - Novartis Investigative Site, Medellín, Antioquia
  - Novartis Investigative Site, Bucaramanga, Colombia
  - Novartis Investigative Site, Medellín, Colombia
  - Novartis Investigative Site, Bogota, Cundinamarca
  - Novartis Investigative Site, Bogotá
- Estonia (4):
  - Novartis Investigative Site, Tartu, Estonia
  - Novartis Investigative Site, Kohtla-Järve
  - Novartis Investigative Site, Tallinn
  - Novartis Investigative Site, Tartu
- Germany (13):
  - Novartis Investigative Site, Bochum, Germany
  - Novartis Investigative Site, Marburg, Germany
  - Novartis Investigative Site, Bad Wörishofen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Darmstadt
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Gauting
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Landsberg
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Lübeck
  - Novartis Investigative Site, Mainz
- Hungary (7):
  - Novartis Investigative Site, Szarvas, Hungary
  - Novartis Investigative Site, Szeged, Hungary
  - Novartis Investigative Site, Győr, HUN
  - Novartis Investigative Site, Százhalombatta, HUN
  - Novartis Investigative Site, Törökbálint, Pest County
  - Novartis Investigative Site, Cegléd
  - Novartis Investigative Site, Gödöllő
- India (12):
  - Novartis Investigative Site, Ahmedabad, Gujarat
  - Novartis Investigative Site, Vadodara, Gujarat
  - Novartis Investigative Site, Bangalore, Karnataka
  - Novartis Investigative Site, Hubli, Karnataka
  - Novartis Investigative Site, Mysore, Karnataka
  - Novartis Investigative Site, Cherthala, Kerala
  - Novartis Investigative Site, Mumbai, Maharashtra
  - Novartis Investigative Site, Nagpur, Maharashtra
  - Novartis Investigative Site, Bikaner, Rajasthan
  - Novartis Investigative Site, Coimbatore, Tamil Nadu
  - Novartis Investigative Site, Hyderabad, Telangana
  - Novartis Investigative Site, Varanasi, Uttar Pradesh
- Italy (5):
  - Novartis Investigative Site, Cassano delle Murge, BA
  - Novartis Investigative Site, Florence, FI
  - Novartis Investigative Site, Genova, Italy
  - Novartis Investigative Site, Fiumicino, RM
  - Novartis Investigative Site, Roma
- Japan (5):
  - Novartis Investigative Site, Chuo Ku, Tokyo
  - Novartis Investigative Site, Chuo-ku, Tokyo
  - Novartis Investigative Site, Setagaya-ku, Tokyo
  - Novartis Investigative Site, Shinjuku-ku, Tokyo
  - Novartis Investigative Site, Toshima-ku, Tokyo
- Latvia (4):
  - Novartis Investigative Site, Jūrmala, LVA
  - Novartis Investigative Site, Riga, LV
  - Novartis Investigative Site, Daugavpils
  - Novartis Investigative Site, Riga
- Novartis Investigative Site, Vilnius, Lithuania
- Malaysia (4):
  - Novartis Investigative Site, Alor Star, Kedah
  - Novartis Investigative Site, Taiping, Perak
  - Novartis Investigative Site, Kuala Terengganu, Terengganu
  - Novartis Investigative Site, Putrajaya
- Peru (4):
  - Novartis Investigative Site, Santiago de Surco, Lima region
  - Novartis Investigative Site, Cusco
  - Novartis Investigative Site, Lima
  - Novartis Investigative Site, Piura
- Philippines (3):
  - Novartis Investigative Site, Iloilo City, Iloilo
  - Novartis Investigative Site, Manila
  - Novartis Investigative Site, Quezon City
- Poland (4):
  - Novartis Investigative Site, Biaystok, Poland
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Grudziądz
  - Novartis Investigative Site, Katowice
- Russia (4):
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Rostov-on-Don
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yekaterinburg
- Slovakia (13):
  - Novartis Investigative Site, Bardejov, Slovak Republic
  - Novartis Investigative Site, Bojnice, Slovak Republic
  - Novartis Investigative Site, Humenné, Slovak Republic
  - Novartis Investigative Site, Liptovský Hrádok, Slovak Republic
  - Novartis Investigative Site, Spišská Nová Ves, Slovak Republic
  - Novartis Investigative Site, Stropkov, Slovak Republic
  - Novartis Investigative Site, Čadca, Slovakia
  - Novartis Investigative Site, Prešov, Slovakia
  - Novartis Investigative Site, Zvolen, Slovakia
  - Novartis Investigative Site, Banská Bystrica, SVK
  - Novartis Investigative Site, Poprad, SVK
  - Novartis Investigative Site, Bratislava
  - Novartis Investigative Site, Sabinov
- South Africa (6):
  - Novartis Investigative Site, Winnie Mandela, Free State
  - Novartis Investigative Site, Middelburg, Mpumalanga
  - Novartis Investigative Site, Belleville, South Africa
  - Novartis Investigative Site, Cape Town, ZAF
  - Novartis Investigative Site, Cape Town
  - Novartis Investigative Site, Panorama
- South Korea (8):
  - Novartis Investigative Site, Anyang-si, Gyeonggi-do
  - Novartis Investigative Site, Bucheon-si, Gyeonggi-do
  - Novartis Investigative Site, Hwaseong-si, Gyeonggi-do
  - Novartis Investigative Site, Suwon, Gyeonggi-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Seoul, Seocho gu
  - Novartis Investigative Site, Busan
  - Novartis Investigative Site, Seoul
- Sweden (3):
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
  - Novartis Investigative Site, Linköping, Östergötland County
- Thailand (3):
  - Novartis Investigative Site, Bangkok, Thailand
  - Novartis Investigative Site, Khon Kaen, THA
  - Novartis Investigative Site, Chiang Mai
- Vietnam (2):
  - Novartis Investigative Site, Ho Chi Minh City, VNM
  - Novartis Investigative Site, Haiphong

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Oba Y, Anwer S, Maduke T, Patel T, Dias S. Effectiveness and tolerability of dual and triple combination inhaler therapies compared with each other and varying doses of inhaled corticosteroids in adolescents and adults with asthma: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2022 Dec 6;12(12):CD013799. doi: 10.1002/14651858.CD013799.pub2. PMID 36472162
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=730
- See also: A Pediatric Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/ppatientsummary/ppatientsummaries?periodicPatientSummaryId=512

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | QMF149 150/80 μg | MF 200 µg
Started | 398 | 404
Full analysis set | 395 | 399
Completed | 394 | 383
Not Completed | 4 | 21
Not completed — Protocol deviation | 3 | 4
Not completed — Adverse Event | 1 | 8
Not completed — Lost to Follow-up | 0 | 1
Not completed — Non-compliance with study treatment | 0 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Subject/guardian decision | 0 | 4
Not completed — Technical problems | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | QMF149 150/80 μg | MF 200 µg | Total
Number analyzed (Participants) | 398 | 404 | 802
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.1 (16.26) | 45.1 (16.27) | 45.6 (16.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 247 | 241 | 488
  Male | 151 | 163 | 314
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 98 | 101 | 199
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 5 | 6
  White | 262 | 265 | 527
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 37 | 33 | 70

OUTCOME MEASURES:

1. Primary Outcome: Trough FEV1
Description: demonstrate the superiority of QMF149 150/80 microgram o.d. (in the evening) delivered via Concept1 compared with MF 200 microgram o.d. (in the evening) delivered via Twisthaler® in terms of trough FEV1 after 12 weeks of treatment in adults and adolescents. Forced Expiratory Volume in 1 second (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured by spirometry.
Time Frame: week 12
Population: The Full Analysis Set (FAS) consisted of all patients in the RAN set who received at least one dose of study treatment. Following the intent-to-treat principle, patients were analyzed according to the treatment they were assigned to at randomization. The FAS was used in the analysis of all efficacy variables.
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QMF149 150/80 μg | MF 200 µg
Number analyzed (Participants) | 395 | 399
Liters | 2.562 (0.0134) | 2.379 (0.0134)
Statistical Analysis 1: Comparison: QMF149 150/80 μg vs MF 200 µg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.182, 95% CI 2-sided [0.148 to 0.217]

2. Secondary Outcome: ACQ-7
Description: ACQ-7 is an asthma control questionnaire (scoring 5 symptoms, FEV1 entered by the investigator and daily rescue bronchodilator use entered by the patient) validated to evaluate different levels of asthma control. the ACQ-7 was used to assess improvements in asthma symptom control. The ACQ-7, a seven-item disease-specific instrument developed and validated to assess asthma control in patients in clinical trials as well as in individuals in clinical practice, was provided to the site. All seven items were then scored on a 7-point Likert scale, with 0 indicating total control and 6 indicating no control. The questions were equally weighted and the total score was the mean of the seven items. The first 6 questions of the ACQ-7 were completed by the patient while the last question (question 7) was completed by the study investigator using spirometry data generated by the spirometry equipment.
Time Frame: week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | QMF149 150/80 μg | MF 200 µg
Number analyzed (Participants) | 395 | 399
Units on a scale | 1.323 (0.0411) | 1.540 (0.0411)
Statistical Analysis 1: Comparison: QMF149 150/80 μg vs MF 200 µg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.218, 95% CI 2-sided [-0.293 to -0.143]

3. Secondary Outcome: Trough FEV1 at Day 2
Description: Forced Expiratory Volume in 1 second (FEV1) is the amount of air which can be forcibly exhaled from the lungs in the first second of a forced exhalation, measured through spirometry testing
Time Frame: Day 2
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QMF149 150/80 μg | MF 200 µg
Number analyzed (Participants) | 395 | 399
Liters | 2.490 (0.0108) | 2.358 (0.0108)
Statistical Analysis 1: Comparison: QMF149 150/80 μg vs MF 200 µg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.132, 95% CI 2-sided [0.105 to 0.158]

4. Secondary Outcome: Pre-dose FEV1 at Week 4
Description: Pre-dose FEV1 is defined as the mean of -45 min and -15 min FEV1 values pre-evening dose
Time Frame: week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QMF149 150/80 μg | MF 200 µg
Number analyzed (Participants) | 395 | 399
Liters | 2.545 (0.0132) | 2.369 (0.0131)
Statistical Analysis 1: Comparison: QMF149 150/80 μg vs MF 200 µg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.176, 95% CI 2-sided [0.145 to 0.207]

5. Secondary Outcome: FVC Over 12 Weeks
Description: FVC is the total amount of air exhaled during the FEV test. Forced Vital Capacity (FVC) and Forced Expiratory Flow between 25% and 75% of FVC (FEF25-75) will be measured
Time Frame: week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | QMF149 150/80 μg | MF 200 µg
Number analyzed (Participants) | 395 | 399
Liters
  Pre dose trough FVC (n=383,379): number analyzed (Participants) | 383 | 379
  Pre dose trough FVC (n=383,379) | 3.453 (0.0169) | 3.353 (0.0169)
  Pre-dose trough FEF25-75% (n=383,379): number analyzed (Participants) | 383 | 379
  Pre-dose trough FEF25-75% (n=383,379) | 2.030 (0.0228) | 1.742 (0.0228)
Statistical Analysis 1: Comparison: QMF149 150/80 μg vs MF 200 µg; Pre-dose trough FVC; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.100, 95% CI 2-sided [0.061 to 0.139]
Statistical Analysis 2: Comparison: QMF149 150/80 μg vs MF 200 µg; Pre-dose trough FEF25-75%; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.288, 95% CI 2-sided [0.231 to 0.345]

6. Secondary Outcome: PEF Over 4 and 12 Weeks
Description: Morning and Evening Peak Expiratory Flow Rate (PEF) will be measured. PEF is the peak expiratory flow, the maximum speed of expiration
Time Frame: week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: L/min
Arm/Group | QMF149 150/80 μg | MF 200 µg
Number analyzed (Participants) | 395 | 399
L/min
  Mean Morning PEF (n=382,382): number analyzed (Participants) | 382 | 382
  Mean Morning PEF (n=382,382) | 31.0 (1.98) | 3.8 (1.97)
  Mean Evening PEF (n=386,386): number analyzed (Participants) | 386 | 386
  Mean Evening PEF (n=386,386) | 26.8 (1.84) | 0.7 (1.84)
Statistical Analysis 1: Comparison: QMF149 150/80 μg vs MF 200 µg; Mean Morning PEF; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 27.2, 95% CI 2-sided [22.1 to 32.4]
Statistical Analysis 2: Comparison: QMF149 150/80 μg vs MF 200 µg; Mean Evening PEF; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 26.1, 95% CI 2-sided [21.0 to 31.2]

7. Secondary Outcome: Percentage of Patients With ACQ-7 MID at Week 12
Description: MID is Minimum Important Difference. ACQ-7 is an asthma control questionnaire (scoring 5 symptoms, FEV1 entered by the investigator and daily rescue bronchodilator use entered by the patient) validated to evaluate different levels of asthma control. Percent of patients achieving the minimal important difference (MID) in ACQ-7 (i.e. at least 0.5 decrease from baseline) will be measured.
Time Frame: week 12
Population: as for outcome 1
Measure: Number; unit: Percentage
Arm/Group | QMF149 150/80 μg | MF 200 µg
Number analyzed (Participants) | 395 | 399
Percentage | 74.7 | 64.9

8. Secondary Outcome: Daily E-diary Over 12 Weeks
Description: Percentage of asthma symptoms free days, the percentage of nights without nighttime awakenings, and the percentage of mornings without symptoms on awakening as recorded by daily electronic Diary (e-Diary) over 12 weeks of treatment
Time Frame: week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | QMF149 150/80 μg | MF 200 µg
Number analyzed (Participants) | 395 | 399
Percentage
  % of nights with no night-time awakenings: number analyzed (Participants) | 384 | 384
  % of nights with no night-time awakenings | 13.4 (1.37) | 8.7 (1.36)
  % of mornings with no symptoms on awakening: number analyzed (Participants) | 384 | 384
  % of mornings with no symptoms on awakening | 14.7 (1.53) | 11.2 (1.53)
  % of asthma symptom-free days: number analyzed (Participants) | 373 | 380
  % of asthma symptom-free days | 17.1 (1.68) | 14.4 (1.65)

9. Secondary Outcome: ACQ-7 at Week 4
Description: ACQ-7 is an asthma control questionnaire (scoring 5 symptoms, FEV1 entered by the investigator and daily rescue bronchodilator use entered by the patient) validated to evaluate different levels of asthma control
Time Frame: week 4
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | QMF149 150/80 μg | MF 200 µg
Number analyzed (Participants) | 395 | 399
Units on a scale | 1.454 (0.0408) | 1.658 (0.0406)
Statistical Analysis 1: Comparison: QMF149 150/80 μg vs MF 200 µg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.204, 95% CI 2-sided [-0.277 to -0.131]

10. Secondary Outcome: Rescue Medication Use Over 12 Weeks
Description: Rescue salbutamol/albuterol usage (mean daily, nighttime and daytime use) from e-Diary recordings over 12 weeks of treatment
Time Frame: week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Number of puffs of rescue medication
Arm/Group | QMF149 150/80 μg | MF 200 µg
Number analyzed (Participants) | 395 | 399
Number of puffs of rescue medication
  Night-time number of puffs of rescue medication: number analyzed (Participants) | 384 | 384
  Night-time number of puffs of rescue medication | -0.26 (0.025) | -0.16 (0.025)
  Daytime number of puffs of rescue medication: number analyzed (Participants) | 388 | 389
  Daytime number of puffs of rescue medication | -0.39 (0.033) | -0.24 (0.032)
Statistical Analysis 1: Comparison: QMF149 150/80 μg vs MF 200 µg; Night-time number of puffs of rescue medication; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.16 to -0.05]
Statistical Analysis 2: Comparison: QMF149 150/80 μg vs MF 200 µg; Daytime number of puffs of rescue medication; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = -0.15, 95% CI 2-sided [-0.22 to -0.08]

11. Secondary Outcome: Percentage of Rescue Medication Free Days Over 12 Weeks
Description: Percentage of rescue medication free days over 12 weeks of treatment period
Time Frame: week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | QMF149 150/80 μg | MF 200 µg
Number analyzed (Participants) | 395 | 399
Percentage | 22.2 (1.81) | 14.1 (1.80)
Statistical Analysis 1: Comparison: QMF149 150/80 μg vs MF 200 µg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 8.1, 95% CI 2-sided [4.3 to 11.8]

12. Secondary Outcome: Quality of Life Assessed by Asthma Quality of Life Questionnaire AQLQ-S 12
Description: The AQLQ is a 32-item disease specific questionnaire designed to measure functional impairments in asthma. Patients are asked to score each item on a 7-point scale based on the experience of last 2 weeks. The overall AQLQ score is the mean response to all 32 questions. Therefore, the possible highest score (better) would be 7 and the lowest (worse) would be 1. Changes in scores of 0.5 to 1.0 are considered clinically meaningful; 1.0 to 1.5 as moderate and > 1.5 as marked clinically important differences for any individual domain or for the overall summary score.
Time Frame: week 12
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Score
Arm/Group | QMF149 150/80 μg | MF 200 µg
Number analyzed (Participants) | 395 | 399
Score | 5.779 (0.0475) | 5.630 (0.0473)
Statistical Analysis 1: Comparison: QMF149 150/80 μg vs MF 200 µg; Test type: Superiority; p < 0.001, Mixed Models Analysis; Mean Difference (Net) = 0.149, 95% CI 2-sided [0.064 to 0.234]

13. Secondary Outcome: Number of Patients With Asthma Exacerbation Over 12 Weeks
Description: The exacerbation categories are: mild, moderate, severe and the combination of moderate or severe. Time to first asthma exacerbation by exacerbation category. Annual rate of asthma exacerbations by exacerbation category.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Number of patients
Arm/Group | QMF149 150/80 μg | MF 200 µg
Number analyzed (Participants) | 395 | 399
Number of patients
  Mild asthma exacerbation | 11 | 29
  Moderate asthma exacerbation | 7 | 23
  Severe asthma exacerbation | 3 | 11
  Moderate or severe asthma exacerbation | 10 | 32

14. Secondary Outcome: The Number of Asthma Exacerbations (Moderate or Severe) Over the 12 Week Treatment Period
Description: Annual incidence rate of asthma exacerbation by severity of exacerbation. The number of asthma exacerbation is used to calculate annual incidence rate. A severe asthma exacerbation is SCS (Systemic Corticosteroids) use ≥3 days and hospitalization or emergency department visit (greater than 24 h) or death due to asthma. A moderate asthma exacerbation is SCS use ≥3 days either as an outpatient or in emergency department visits (less than or equal to 24 h). Worsening of asthma not requiring more than 3 days of SCS or hospitalization/emergency room will be considered mild asthma exacerbations
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Number of exacerbation
Arm/Group | QMF149 150/80 μg | MF 200 µg
Number analyzed (Participants) | 395 | 399
Number of exacerbation
  Moderate or severe asthma exacerbation: number analyzed (Participants) | 394 | 397
  Moderate or severe asthma exacerbation | 0.08 | 0.31
  All (mild, moderate, severe) asthma exacerbation: number analyzed (Participants) | 394 | 397
  All (mild, moderate, severe) asthma exacerbation | 0.20 | 0.67

15. Secondary Outcome: Number of Patients With First Asthma Exacerbations (Moderate or Severe) Over the 12 Week Treatment Period
Description: The annual rate of asthma exacerbations were analyzed using a generalized linear model.
Time Frame: Week 12
Population: as for outcome 1
Measure: Number; unit: Count of participants
Arm/Group | QMF149 150/80 μg | MF 200 µg
Number analyzed (Participants) | 395 | 399
Count of participants | 10 | 32
Statistical Analysis 1: Comparison: QMF149 150/80 μg vs MF 200 µg; Test type: Superiority; p < 0.001, Regression, Cox; Hazard Ratio (HR) = 0.29, 95% CI 2-sided [0.14 to 0.59]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: AE additional description
Groups:
- QMF149 150/80: QMF149 150/80 microgram o.d. delivered via Concept1
- MF 200: MF 200 microgram o.d. delivered via Twisthaler®
Arm/Group | QMF149 150/80 | MF 200
All-Cause Mortality (participants affected / at risk) | 0/396 | 0/399
Serious Adverse Events (participants affected / at risk) | 5/396 | 7/399
Other Adverse Events (participants affected / at risk) | 69/396 | 106/399
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | QMF149 150/80 (N=396) | MF 200 (N=399)
Appendix disorder (Gastrointestinal disorders) | 0 | 1
Dental cyst (Gastrointestinal disorders) | 1 | 0
Autoimmune hepatitis (Hepatobiliary disorders) | 0 | 1
Abscess oral (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 0 | 1
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | QMF149 150/80 (N=396) | MF 200 (N=399)
Bronchitis (Infections and infestations) | 1 | 5
Influenza (Infections and infestations) | 4 | 4
Nasopharyngitis (Infections and infestations) | 17 | 19
Pharyngitis (Infections and infestations) | 5 | 2
Sinusitis (Infections and infestations) | 5 | 5
Upper respiratory tract infection (Infections and infestations) | 4 | 10
Viral upper respiratory tract infection (Infections and infestations) | 1 | 5
Overdose (Injury, poisoning and procedural complications) | 5 | 10
Headache (Nervous system disorders) | 4 | 9
Asthma (Respiratory, thoracic and mediastinal disorders) | 20 | 60
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 5 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 4
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety

DOCUMENTS (2):
  • Study Protocol (2018-03-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT02892344/Prot_000.pdf
  • Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/44/NCT02892344/SAP_001.pdf